# Official Title: Prediction of Recipient Renal Function in Living Donor Kidney Transplantation Using Baseline Characteristics and Donor Renal Volume

**ClinicalTrials.gov NCT Number:** 

**Document Date: December 2, 2024** 

### 1. Purpose and Background

Kidney transplantation is the definitive treatment for end-stage renal disease (ESRD). Accurately predicting early post-transplant kidney function is critical for patient management and improving long-term outcomes. This study aims to develop a machine learning-based predictive model using baseline characteristics of recipients and donors, with a focus on donor kidney volume, to predict the lowest serum creatinine level within one year post-transplant.

#### 2. Study Design

- **Study Type**: Retrospective Cohort Study
- **Duration**: January 2006- March 2023
- **Setting**: Multicenter study conducted at Seoul National University Hospital, Severance Hospital, and Bundang Seoul National University Hospital.
- Participants: Living-donor kidney transplant recipients and their corresponding donors.

## 3. Eligibility Criteria

#### **Inclusion Criteria:**

• Living-donor kidney transplant recipients and donors from the above centers.

#### **Exclusion Criteria:**

- Recipients or donors with follow-up duration less than 1 year.
- Recipients younger than 18 years old.
- Re-transplantation cases or recipients with simultaneous multi-organ transplantation.

## 4. Data Collection and Management Plan

- Data was retrieved from hospital records and centralized in a unified dataset.
- Variables included demographic data, donor kidney volume (total and cortex), recipient-donor compatibility, and baseline laboratory data.

## 5. Primary and Secondary Outcomes

- **Primary Outcome**: Lowest serum creatinine level within one year post-transplant.
- **Secondary Outcomes**: Predictive performance metrics (MAE, RMSE, R<sup>3</sup>), donor kidney volume correlations with recipient eGFR, and subgroup analyses by donor type.

## 6. Statistical Analysis

#### 6.1 Statistical Software

All statistical analyses and data preprocessing will be conducted using the following software tools:

# 1. R Software (Version 4.4.1):

 Primary software for statistical analyses, including descriptive statistics, hypothesis testing, and data visualization.

# 2. Python (Version 3.9):

o Used for developing and validating machine learning models.

#### **6.2 Predictive Model Development**

## **Algorithms Used:**

- Multiple Linear Regression (with and without variable selection)
- Elastic Net
- Generalized Additive Model (GAM)
- Random Forest
- Gradient Boosting (XGBoost)

## **Variable Selection Methods:**

- Multiple Linear Regression: AIC-based stepwise selection.
- Elastic Net: LASSO regularization.
- GAM: Cross-validation for smoothing parameter selection.

Tree-based models (Random Forest, Gradient Boosting, XGBoost): Feature importance evaluation based on cross-validation.

# **Hyperparameter Tuning:**

Grid search with 5-fold cross-validation will be used to optimize hyperparameters for machine learning models.

#### 6.3 Model Evaluation

#### **Performance Metrics:**

1. Mean Absolute Error (MAE):

$$MAE = \frac{1}{n} \sum_{i=1}^{n} |y_i - \hat{y}_i|$$

y<sub>i</sub>: Actual value

 $\hat{y}_i$ : Predicted value

n=Number of observations

2. Root Mean Square Error (RMSE):

RMSE= 
$$\sqrt{\frac{1}{n}\sum_{i=1}^{n}(y_{i}-\hat{y}_{i})^{2}}$$

y<sub>i</sub>: Actual value

 $\hat{y}_i$ : Predicted value n=Number of observations

3. R-squared (R<sup>2</sup>):

$$R^{2} = 1 - \frac{SS_{res}}{SS_{tot}}$$

 $SS_{res} = \sum_{i=1}^{n} (y_i - \hat{y}_i)^2$ : Residual Sum of Square

SS<sub>tot</sub>= $\sum_{i=1}^{n} |y_i - \bar{y}_i|$ : Total Sum of Squares

#### **Internal Validation**:

Models will be evaluated using the internal validation set for all performance metrics.

## **External Validation:**

• The final model will be tested on the external validation set to assess generalizability.

# **6.4 Subgroup Analysis**

 Subgroups based on recipient characteristics (e.g., sex, age, baseline BMI) and donor variables (e.g., kidney volume) will be analyzed to evaluate heterogeneity in model performance.

# **6.5 Feature Importance Analysis**

• Feature importance scores will be derived from tree-based models (Random Forest, XGBoost) to identify the most influential predictive variables.

## 7. Ethical Considerations

- Approved by the SNUH Institutional Review Board (IRB No. H-2205-051-1322).
- Study participants provided informed consent for data usage.